CLINICAL TRIAL: NCT03895411
Title: Multicenter Clinical Study of Therapeutic Effect of Sotalol on Children With Arrhythmia (Paroxysmal Supraventricular Tachycardia, Paroxysmal Atrial Tachycardia, Ventricular Tachycardia, Idiopathic Ventricular Tachycardia, Premature Ventricular Contraction ) in Children Aged From 0d to 14 Yrs
Brief Title: Efficacy and Safety of Sotalol in Children With Arrhythmia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Hong Wang, Professor, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJEX001
Record Dates: First submitted 2019-03-25; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Sotalol; Propafenone; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sotalol (Experimental): Oral sotalol 2.5mg/kg/time, per 12h. Combination therapy: betaloc
  Interventions: Drug: sotalol; Drug: betaloc
- Propafenone (Active Comparator): Oral Propafenone 5mg/kg/time, pre 8h Combination therapy: betaloc
  Interventions: Drug: Propafenone; Drug: betaloc

INTERVENTIONS:
Drug: sotalol — Oral sotalol 2.5mg/kg/time, per 12h
  Arms: Sotalol
Drug: Propafenone — Oral Propafenone 5mg/kg/time, pre 8h
  Arms: Propafenone
Drug: betaloc — Oral betaloc 0.5mg/kg/time ,pre 12h

SUMMARY:
This study aims to investigate the efficacy and safety of oral sotalol alone or combination with other anti-arrhythmic medicines in the treatment of arrhythmias in children. The study will regularly monitor the Holter, electrocardiogram (ECG), Echocardiography (Echo), blood routine, urine routine, serum ion, liver and kidney function, troponin I, hypersensitive troponin T, N-terminal pro-brain natriuretic peptide (NT pro-BNP), etc, before and after receive sotalol therapy. Compare the degree of arrhythmia improvement in patients and the side effects after oral sotalol.

DETAILED DESCRIPTION:
Monitoring the Holter, ECG, Echocardiography , blood routine, urine routine, serum ion, liver and kidney function, troponin I, hypersensitive troponin T, NT pro-BNP beforehand. Eligible patients should stop all anti-arrhythmia drugs and digitalis, tricyclic antidepressants, beta blockers or calcium antagonists for at least 5 half-lives, and then do Holter. Randomly grouped. Judging the results according to the situation before and after oral sotalol.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0 day to 14 year-old
2. Diagnosis of tachycardia (paroxysmal supraventricular tachycardia, paroxysmal atrial tachycardia, ventricular tachycardia, idiopathic ventricular tachycardia, premature ventricular contraction) and had an episode within 3 months; Premature Ventricular Contractions (PVC) (total 10000 times/d, or>5000 times/d with multiple source PVC, or total > 3000 times/d but with paired PVC+ multiple source PVC, or ventricular tachycardia);
3. Although PVC≤ 10000 times/d, but there are obvious symptoms such as palpitation, chest tightness, fatigue, dizziness and other symptoms that need improvement.
4. Signed informed consent before the trial
5. Good compliance

Exclusion Criteria:

1. Heart failure that is ineffective in conventional treatment;
2. Left ventricular ejection fraction (LVEF) ≤ 50%;
3. Suffering from bronchial asthma;
4. Resting sinus heart rate (HR) in newborns <90 bpm; -8 yrs <80 bpm; ≥ 8 yrs <60 bpm;
5. Corrected QT Interval (QTc) ≥ 450ms;
6. II ° -III ° atrioventricular block (AVB);
7. Severe liver, renal dysfunction, acute myocardial infarction, acute myocarditis, electrolyte imbalance have not been corrected;
8. The child has undergone major surgery in the past 4 weeks;
9. The child has participated in other clinical trials in the past 4 weeks;
10. The child has digestive, nervous, circulatory, kidney or liver disease

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
QT interval of ECG | 1 week
QT interval of ECG | 3 month

SECONDARY OUTCOMES:
Blood pressure | 1 week, 3 month
Red Blood Cell (RBC) | 1 week, 3 month
  The indicator is obtained through blood routine.
Wed Blood Cell (WBC) | 1 week, 3 month
  The indicator is obtained through blood routine.
Hemoglobin | 1 week, 3 month
  The indicator is obtained through blood routine.
Platelet | 1 week, 3 month
  The indicator is obtained through blood routine.
Albumin | 1 week, 3 month
  The indicator is obtained through liver function test.
Alanine aminotransferase (ALT) | 1 week, 3 month
  The indicator is obtained through liver function test.
Aspertate aminotransferase (AST) | 1 week, 3 month
  The indicator is obtained through liver function test.
Creatinine | 1 week, 3 month
  The indicator is obtained through kidney function test.

CONTACTS AND LOCATIONS:
Locations (1):
- Shenjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided
Dear Sir/Madam Our study receives a grant from China Ministry of Science and Technology. We cannot decide whether the data could be shared. Hope you can understand.